CLINICAL TRIAL: NCT01899768
Title: A Randomised, Double-Blind (Sponsor-Unblind), Placebo Controlled, Cross-Over Study to Investigate the Efficacy, Effect on Cough Reflex Sensitivity, Safety, Tolerability and Pharmacokinetics of Inhaled GSK2339345 in Patients With Chronic Idiopathic Cough Using an Aqueous Droplet Inhaler
Brief Title: GSK2339345 Hypertussive Challenge Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: North West Lung Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 117270
Record Dates: First submitted 2013-07-11; First posted 2013-07-15 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-02

CONDITIONS: Cough
Keywords: efficacy; hypertussive challenge; voltage gated sodium channels (VGSC); anaesthesia; Safety and tolerability; capsaicin challenge; cough; citric acid challenge; pharmacokinetics
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A (Experimental): Subjects will receive treatment A (placebo) or treatment B (GSK2339345) in 3 visits of part A (one treatment per visit) in one of the following four sequences: ABA, ABB, BAA, and BAB.
  Interventions: Drug: GSK2339345; Drug: Placebo
- Part B (Experimental): Subjects will receive treatment A or treatment B in 2 visits of part B (one treatment per visit) in one of the following two sequences: AB and BA. Subjects will then orally inhale 10 microliter (mcL) of a capsaicin solution of strength ranging from 0.49 micromolar (mcM) to 1000 mcM, which will be administered using a breath activated dosimeter approximately 5 minutes post-dosing with treatment A or B at Visits 4 and 5.
  Interventions: Drug: GSK2339345; Drug: Placebo
- Part C (Experimental): Subjects will receive treatment A or treatment B in 2 visits of part C (one treatment per visit) in one of the following two sequences: AB and BA. Subjects will then orally inhale 10 mcL of a citric acid solution of strength ranging from 0.03 to 4.0 M, which will be administered using a breath activated dosimeter approximately 5 minutes post-dosing with treatment A or B at Visits 6 and 7.
  Interventions: Drug: GSK2339345; Drug: Placebo

INTERVENTIONS:
Drug: GSK2339345 — Clear colorless solution in clear glass vial for oral inhalation via aqueous droplet inhaler with unit dose strength of 1000 microgram (mcg) inhaled in two actuations.
Drug: Placebo — Clear colorless solution of 0.9% sodium chloride for oral inhalation via aqueous droplet inhaler inhaled in two actuations.

SUMMARY:
This study is designed to evaluate the effect of GSK2339345 relative to placebo on the number of coughs in patients with Chronic Idiopathic Cough (CIC) administered by an Aqueous Droplet Inhaler (ADI). The primary aim is to investigate the efficacy of GSK2339345 on reducing objective cough frequency in CIC patients. The secondary aim of this study is to investigate the efficacy of GSK2339345 in inhibiting a hypertussive cough response elicited by capsaicin and citric acid in CIC patients which have a hyperresponsive cough reflex.

Following the screening visit, all eligible subjects will attend the unit for dosing at Visits 1-7. At Visits 1, 2 and 3 (Part A of the study), subjects will receive two doses of either GSK2339345 or placebo, 4 hours apart and will undergo 8 hours of cough monitoring. At Visits 4 and 5 (Part B of the study) and Visits 6 and 7 (Part C of the study), subjects will be administered a single dose of either GSK2339345 or placebo. Subjects will then undergo capsaicin (Part B) or citric acid (Part C) tussive challenge and will undergo cough monitoring for 1 hour post dose.

The maximum study duration will be approximately 11 weeks, including 3 weeks screening and 2 weeks follow-up. Approximately 30 patients will be randomised into the study, such that approximately 24 patients complete dosing and critical assessments.

ELIGIBILITY:
Inclusion Criteria

* Chronic Idiopathic Cough patients according to the criteria listed below, determined by a responsible and experienced physician, based on a medical evaluation: Idiopathic cough defined as chronic cough resistant to treatment targeted at potential triggers. Chronic cough defined as cough lasting for more than 8 weeks.
* A patient with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male/females aged >=18 years old, at the time of signing the informed consent.
* Non-smoker for at least 6 months with a cumulative history of <= 10 pack years. Pack years = (No. of cigarettes smoked/day/20) x (No. of years smoked).
* Body weight >= 50 kilograms.
* A female subject is eligible to participate if she is of; Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone > 40 milli international unit/milliliter (mL) and estradiol < 40 picogram/ml (<147 picomoles/Liter [L]) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2 to4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.

Child-bearing potential with negative pregnancy test as determined by serum human chorionic gonadotropin test at screening or prior to dosing and Agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow up visit or has only same-sex partners, when this is her preferred and usual lifestyle.

* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods. This criterion must be followed from the time of the first dose of study medication until the follow up visit.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Aspartate amino transferase and alanine amino transferase < 2xupper limit of normal (ULN); alkaline phosphatase and bilirubin <= 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on averaged QT interval corrected (QTc) values of triplicate electrocardiograms (ECGs) obtained over a brief recording period: QTc using Fridericia's formula (QTcF) < 450 millisecond.
* A 24 hour Holter ECG at screening that demonstrates no clinically significant abnormalities or finding that could interfere with interpretation of the study results, when assessed by an appropriately trained and experienced reviewer.

Exclusion Criteria Based Upon Medical Histories

* Subjects who have evidence of current asthma, as confirmed by the Investigator or designee.
* Subjects with any clinically significant respiratory condition or lung pathology that could cause cough (apart from chronic idiopathic cough).
* Known lung cancer or other active malignancy, or history of.
* Subjects with current or a chronic history of cardiovascular disease (including uncontrolled hypertension, ischemic heart disease, angina, myocardial infarct, congestive heart failure, and stroke).
* Subjects with current central nervous system / peripheral nervous system conditions e.g. epilepsy and myasthenia gravis.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Any subject with a respiratory tract infection within 4 weeks of screening.
* Radiological imaging prior to the study, including chest X-rays, that have shown any evidence of clinically significant lung disease, as judged by the Investigator or designee.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Any subject who has a history of an allergic reaction to a local anesthetic. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation.
* Any subject who has a known hypersensitivity to capsaicin or citric acid. Exclusion Criteria Based Upon Diagnostic Assessment
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Any subject who, upon oropharyngeal examination, is deemed by the Investigator to be unsuitable for oropharyngeal sensation assessments. This includes any injuries to the mucosa of the mouth or pharynx that could potentially increase systemic absorption e.g. oropharyngeal candidiasis.
* FEV1 less than 80% of the predicted normal value prior to first dosing of the study
* Any subject who does not reach C5 following an oral inhalation of capsaicin at a dose level of 250 micromolar at screening.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A positive pre-study drug/alcohol screen. Other Exclusion Criteria
* Subjects who are unable to use the inhaler satisfactorily.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Belfast

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 117270 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 117270 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117270 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 117270 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117270 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117270 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 117270 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All eligible participants (par.) received treatment of either GSK2339345 or placebo at each visit in Parts A (Visits 1-3), B (Visits 4 and 5) and Part C (Visits 6 and 7).
Groups:
- GSK2339345 1000 µg: Participants received two doses of either GSK2339345 1000 µg or matching placebo as a solution administered via an ADI with a four hour dosing interval at 3 visits (one treatment per visit) in Part A and a single dose at 2 visits (one treatment per visit) in Part B and C. Dose 1 was administered on each treatment day at the same time each morning throughout all of Parts A, B and C. The follow-up of each participant occurred 3-14 days after the last dose. There was a washout of 48 hours to 7 days between visits. Additionally, 5 minutes after the administration of placebo or GSK2339345 at each visit period in Part B and C, participants received an oral inhalation of 10 microliter (µL) of a capsaicin solution at each visit in Part B and 10 µL of a citric acid solution at each visit of Part C. The strength of capsaicin solution ranged from 0.49 to 1000 micromolar (µM) and the citric acid solution strength ranged from 0.03 to 4.0 molar.
Period: Part A
Arm/Group | GSK2339345 1000 µg
Started | 16
Completed | 13
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Period: Part B
Arm/Group | GSK2339345 1000 µg
Started | 13
Completed | 11
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Period: Part C
Arm/Group | GSK2339345 1000 µg
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK2339345 1000 µg/Placebo: Participants received two doses of either GSK2339345 1000 µg or matching placebo as a solution administered via an ADI with a four hour dosing interval at 3 visits (one treatment per visit) in Part A and a single dose at 2 visits (one treatment per visit) in Part B and C. Dose 1 was administered on each treatment day at the same time each morning throughout all of Parts A, B and C. The follow-up of each participant occurred 3-14 days after the last dose. There was a washout of 48 hours to 7 days between visits. Additionally, 5 minutes after the administration of placebo or GSK2339345 at each visit period in Part B and C, participants received an oral inhalation of 10 µL of a capsaicin solution at each visit in Part B and 10 µL of a citric acid solution at each visit of Part C. The strength of capsaicin solution ranged from 0.49 to 1000 µM and the citric acid solution strength ranged from 0.03 to 4.0 molar.
Arm/Group | GSK2339345 1000 µg/Placebo
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.7 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 3
Race/Ethnicity, Customized [Number; unit: participants]
  White - White/Caucasian/European Heritage | 16

OUTCOME MEASURES:

1. Primary Outcome: Total Cough Count Over 8 Hours at Visits 1, 2 and 3 (Part A)
Description: Total cough count (8 hours [hr] of recording) was conducted at Visits 1, 2 and 3. Coughs were counted by a cough monitor fitted to the participants for 8 hr post Dose 1. The cough count was calculated as the sum of two four hour cough count totals, with the first four hours starting from the time of the first dose and the second four hours starting at the time of the second dose. The cough counts were sum-up by the treatments received by the participants. Number of coughs in 8 hr period was loge transformed and used for the analysis. Values were imputed pro-rata if 8 hr epoch was less than 8 hr. Mean of the total cough counts recorded post dose of every treatment i.e. placebo or GSK2339345 1000mcg was reported.
Time Frame: Up to 8 hours post-dose at Visits 1, 2 and 3 (Part A)
Population: All Subjects Population comprised of all participants who receive at least one dose of study medication. Only participants with at least one 8 hr cough count were analyzed.
Measure: Geometric Mean (Standard Error); unit: cough count
Groups:
- Placebo: Participants received two doses of placebo as a solution administered via an ADI with a four hour dosing interval, either at one or two visits in Part A (Visits 1, 2 and 3) and a single dose at one of the 2 visits in Parts B (Visits 4 and 5) and Part C (Visits 6 and 7). Dose 1 was administered on each treatment day at the same time each morning throughout all of Parts A, B and C. The follow-up of each participant occurred 3-14 days after the last dose. There was a washout of 48 hours to 7 days between visits. Additionally, 5 minutes after the administration of placebo at each visit in Part B and C, participants received an oral inhalation of 10 µL of a capsaicin solution at each visit in Part B and 10 µL of a citric acid solution at each visit in Part C. The strength of capsaicin solution ranged from 0.49 to 1000 µM and the citric acid solution strength ranged from 0.03 to 4.0 molar.
- GSK2339345 1000 Microgram (mcg): Participants received two doses of GSK2339345 1000 mcg via an ADI with a four hour dosing interval, either at one or two visits in Part A (Visits 1, 2 and 3) and a single dose at one of the 2 visits in Parts B (Visits 4 and 5) and Part C (Visits 6 and 7). Dose 1 was administered on each treatment day at the same time each morning throughout all of Parts A, B and C. The follow-up of each participant occurred 3-14 days after the last dose. There was a washout of 48 hours to 7 days between visits. Additionally, 5 minutes after the administration of placebo at each visit in Part B and C, participants received an oral inhalation of 10 µL of a capsaicin solution at each visit in Part B and 10 µL of a citric acid solution at each visit in Part C. The strength of capsaicin solution ranged from 0.49 to 1000 µM and the citric acid solution strength ranged from 0.03 to 4.0 molar.
Arm/Group | Placebo | GSK2339345 1000 Microgram (mcg)
Number analyzed (Participants) | 14 | 14
cough count | 152.7 (0.226) | 192.5 (0.226)
Statistical Analysis 1: Comparison: Placebo vs GSK2339345 1000 Microgram (mcg); Test type: Superiority or Other; Ratio of adjusted geometric mean = 1.26, 90% CI 2-sided [1.10 to 1.44] — Ratio of adjusted geometric means = GSK2339345/Placebo

2. Primary Outcome: Total Cough Count Excluding Transient Coughs Over 8 Hours at Visits 1, 2 and 3 (Part A)
Description: Total cough count (8 hr of recording) was conducted at Visits 1, 2 and 3. Coughs were counted by a cough monitor fitted to the participants for 8 hr post Dose 1. The cough count was calculated as the sum of two four hour cough count totals, with the first 4-hrs starting from the time of the first dose and the second four hours starting at the time of the second dose. The cough counts were sum-up by the treatments received by the participants. Transient cough was the total number of coughs experienced in the two mins from the start of the first inhalation of a dose. Number of coughs excluding transient cough in 8 hr period was loge transformed and used for the analysis. Values were imputed pro-rata if 8 hr epoch was less than 8 hr. Mean of the total cough counts excluding transient cough recorded post dose of every treatment i.e. placebo or GSK2339345 1000 mcg was reported.
Time Frame: Up to 8 hours post-dose at Visits 1, 2 and 3 (Part A)
Population: All Subjects Population. Only participants with at least one 8 hr cough count were analyzed.
Measure: Geometric Mean (Standard Error); unit: Cough count
Groups:
- GSK2339345 1000 µg: Participants received two doses of GSK2339345 1000 µg via an ADI with a four hour dosing interval, either at one or two visits in Part A (Visits 1, 2 and 3) and a single dose at one of the 2 visits in Parts B (Visits 4 and 5) and Part C (Visits 6 and 7). Dose 1 was administered on each treatment day at the same time each morning throughout all of Parts A, B and C. The follow-up of each participant occurred 3-14 days after the last dose. There was a washout of 48 hours to 7 days between visits. Additionally, 5 minutes after the administration of placebo at each visit in Part B and C, participants received an oral inhalation of 10 µL of a capsaicin solution at each visit in Part B and 10 µL of a citric acid solution at each visit in Part C. The strength of capsaicin solution ranged from 0.49 to 1000 µM and the citric acid solution strength ranged from 0.03 to 4.0 molar.
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 14 | 14
Cough count | 151.5 (0.237) | 153.9 (0.237)
Statistical Analysis 1: Comparison: Placebo vs GSK2339345 1000 µg; Test type: Superiority or Other; Ratio of adjusted geometric mean = 1.02, 90% CI 2-sided [0.87 to 1.19] — Ratio of adjusted geometric means = GSK2339345/Placebo

3. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Any Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, or is an important medical events that jeopardize the participants or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition, or a drug-induced liver injury.
Time Frame: From the start of study treatment and until the follow-up contact (up to 8 Weeks)
Population: All Subjects Population
Measure: Number; unit: participants
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
participants
  Any AE | 10 | 5
  Any SAE | 0 | 0

4. Secondary Outcome: Mean Systolic Blood Pressure and Diastolic Blood Pressure at the Indicated Time Points in Parts A, B and C
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) measurements were obtained at following time points: pre-dose, 5 minutes (min), 15 min (only in Part A), 30 min, and 1 hr after first administration (FA) and second administration (SA) in Part A and each dose administration of Parts B and C. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. Pre-Dose is the average (avg) of the triplicate readings taken at the pre-dose assessment.
Time Frame: Pre-dose, 5 min, 15 min (only in Part A), 30 min, and 1 hr post each dose administered in Parts A, B and C (up to 8 weeks)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
Millimeter of mercury (mmHg)
  SBP, Part A, FA, Dose 1, avg Pre-dose, n=16, 14 | 126.1 (14.09) | 123.3 (15.02)
  SBP, Part A, FA, Dose 1, 5 min, n=16, 14 | 125.5 (14.37) | 130.2 (17.16)
  SBP, Part A, FA, Dose 1, 15 min, n=16, 14 | 125.3 (14.06) | 124.1 (14.44)
  SBP, Part A, FA, Dose 1, 30 min, n=16, 14 | 125.6 (14.12) | 124.1 (17.67)
  SBP, Part A, FA, Dose 1, 1 hr, n=16, 14 | 126.1 (15.66) | 123.6 (13.74)
  SBP, Part A, FA, Dose 2 avg Pre-dose, n=16, 14 | 117.8 (10.95) | 119.5 (11.42)
  SBP, Part A, FA, Dose 2, 5 min, n=15, 14 | 120.6 (13.21) | 128.1 (18.58)
  SBP, Part A, FA, Dose 2, 15 min, n=15, 14 | 120.7 (12.96) | 123.0 (16.15)
  SBP, Part A, FA, Dose 2, 30 min, n=15, 14 | 120.8 (11.97) | 118.2 (12.91)
  SBP, Part A, FA, Dose 2, 1hr, n=15, 14 | 124.5 (13.68) | 121.5 (11.31)
  SBP, Part A, SA, Dose 1, avg Pre-dose, n=7, 7 | 130.8 (15.43) | 121.2 (8.25)
  SBP, Part A, SA, Dose 1, 5 min, n=7, 7 | 127.7 (16.23) | 124.1 (11.17)
  SBP, Part A, SA, Dose 1, 15 min, n=7, 7 | 125.1 (22.35) | 117.9 (9.74)
  SBP, Part A, SA, Dose 1, 30 min, n=7, 7 | 128.0 (18.83) | 119.3 (10.21)
  SBP, Part A, SA, Dose 1, 1 hr, n=7, 7 | 134.4 (17.82) | 122.4 (13.13)
  SBP, Part A, SA, Dose 2 avg Pre-dose, n=7, 7 | 125.0 (11.95) | 112.4 (8.54)
  SBP, Part A, SA, Dose 2, 5 min, n=7, 7 | 125.4 (16.29) | 118.1 (9.32)
  SBP, Part A, SA, Dose 2, 15 min, n=7, 7 | 118.9 (12.40) | 112.4 (9.71)
  SBP, Part A, SA, Dose 2, 30 min, n=7, 7 | 119.0 (11.72) | 116.3 (10.37)
  SBP, Part A, SA, Dose 2, 1hr, n=7, 7 | 129.9 (19.27) | 121.4 (15.09)
  SBP, Part B, avg Pre-dose, n=10, 11 | 119.2 (11.69) | 124.0 (10.42)
  SBP, Part B, 5 min, n=10, 11 | 119.6 (11.24) | 123.9 (13.88)
  SBP, Part B, 15 min, n=10, 11 | 121.5 (15.23) | 118.7 (10.86)
  SBP, Part B, 1 hr, n=10, 11 | 124.2 (17.00) | 125.5 (12.89)
  SBP, Part C, avg Pre-dose, n=9, 9 | 125.2 (11.37) | 123.0 (12.28)
  SBP, Part C, 5 min, n=9, 9 | 125.6 (14.75) | 129.3 (12.70)
  SBP, Part C, 15 min, n=9, 9 | 121.6 (12.24) | 124.1 (13.18)
  SBP, Part C, 1hr, n=9, 9 | 127.1 (15.34) | 135.9 (21.77)
  DBP, Part A, FA, Dose 1, avg Pre-dose, n=16, 14 | 68.8 (7.23) | 69.1 (4.61)
  DBP, Part A, FA, Dose 1, 5 min, n=16, 14 | 72.3 (6.88) | 71.6 (5.33)
  DBP, Part A, FA, Dose 1, 15 min, n=16, 14 | 69.6 (7.80) | 70.6 (6.20)
  DBP, Part A, FA, Dose 1, 30 min, n=16, 14 | 71.6 (10.03) | 69.5 (7.34)
  DBP, Part A, FA, Dose 1, 1 hr, n=16, 14 | 70.9 (7.53) | 69.9 (5.14)
  DBP, Part A, FA, Dose 2 avg Pre-dose, n=16, 14 | 64.6 (5.70) | 65.2 (6.55)
  DBP, Part A, FA, Dose 2, 5 min, n=15, 14 | 66.3 (7.69) | 66.4 (7.69)
  DBP, Part A, FA, Dose 2, 15 min, n=15, 14 | 65.5 (7.90) | 66.1 (8.02)
  DBP, Part A, FA, Dose 2, 30 min, n=15, 14 | 66.7 (7.21) | 67.1 (6.95)
  DBP, Part A, FA, Dose 2, 1hr, n=15, 14 | 68.4 (6.46) | 69.6 (8.78)
  DBP, Part A, SA, Dose 1, avg Pre-dose, n=7, 7 | 70.2 (5.74) | 70.6 (7.93)
  DBP, Part A, SA, Dose 1, 5 min, n=7, 7 | 68.9 (6.20) | 67.9 (4.45)
  DBP, Part A, SA, Dose 1, 15 min, n=7, 7 | 68.6 (4.54) | 67.3 (6.37)
  DBP, Part A, SA, Dose 1, 30 min, n=7, 7 | 67.0 (5.72) | 68.7 (3.30)
  DBP, Part A, SA, Dose 1, 1 hr, n=7, 7 | 72.4 (7.00) | 69.1 (6.49)
  DBP, Part A, SA, Dose 2 avg Pre-dose, n=7, 7 | 67.3 (5.95) | 63.3 (2.89)
  DBP, Part A, SA, Dose 2, 5 min, n=7, 7 | 65.1 (5.98) | 67.0 (4.97)
  DBP, Part A, SA, Dose 2, 15 min, n=7, 7 | 64.4 (5.91) | 64.0 (4.97)
  DBP, Part A, SA, Dose 2, 30 min, n=7, 7 | 63.4 (6.73) | 66.3 (5.25)
  DBP, Part A, SA, Dose 2, 1hr, n=7, 7 | 69.1 (7.90) | 71.3 (5.82)
  DBP, Part B, avg Pre-dose, n=10, 11 | 63.9 (4.74) | 67.3 (4.29)
  DBP, Part B, 5 min, n=10, 11 | 63.9 (3.31) | 66.5 (3.67)
  DBP, Part B, 15 min, n=10, 11 | 64.9 (6.51) | 66.2 (6.00)
  DBP, Part B, 1 hr, n=10, 11 | 64.3 (6.99) | 66.2 (2.82)
  DBP, Part C, avg Pre-dose, n=9, 9 | 64.9 (5.50) | 68.0 (8.68)
  DBP, Part C, 5 min, n=9, 9 | 68.0 (7.37) | 65.6 (5.98)
  DBP, Part C, 15 min, n=9, 9 | 65.7 (4.03) | 65.7 (7.09)
  DBP, Part C, 1hr, n=9, 9 | 65.4 (6.31) | 67.7 (6.71)

5. Secondary Outcome: Mean Heart Rate at the Indicated Time Points in Parts A, B and C
Description: Heart rate measurements were obtained at following time points: pre-dose, 5 min, 15 min (only in Part A), 30 min, and 1 hr after FA and SA in Part A and each dose administration in Parts B and C. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. Pre-Dose is the average of the triplicate readings taken at the pre-dose assessment.
Time Frame: Pre-dose, 5 min, 15 min (only in Part A), 30 min, and 1 hr after each dose administered in Parts A, B and C (up to 8 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
Beats per minute
  Part A, FA, Dose 1, avg Pre-dose, n=16, 14 | 68.6 (7.44) | 66.3 (9.90)
  Part A, FA, Dose 1, 5 min, n=16, 14 | 64.1 (7.50) | 66.5 (10.06)
  Part A, FA, Dose 1, 15 min, n=16, 14 | 64.0 (6.41) | 64.9 (9.57)
  Part A, FA, Dose 1, 30 min, n=16, 14 | 64.1 (10.60) | 61.8 (8.75)
  Part A, FA, Dose 1, 1 hr, n=16, 14 | 62.6 (7.70) | 61.6 (7.88)
  Part A, FA, Dose 2 avg Pre-dose, n=16, 14 | 72.6 (9.27) | 69.4 (11.82)
  Part A, FA, Dose 2, 5 min, n=16, 14 | 69.9 (7.29) | 69.7 (12.02)
  Part A, FA, Dose 2, 15 min, n=16, 14 | 69.0 (7.80) | 68.3 (9.52)
  Part A, FA, Dose 2, 30 min, n=16, 14 | 68.6 (9.25) | 68.5 (13.39)
  Part A, FA, Dose 2, 1hr, n=16, 14 | 68.5 (8.30) | 67.6 (11.57)
  Part A, SA, Dose 1, avg Pre-dose, n=7, 7 | 66.8 (12.80) | 69.6 (8.33)
  Part A, SA, Dose 1, 5 min, n=7, 7 | 61.3 (8.90) | 65.4 (8.08)
  Part A, SA, Dose 1, 15 min, n=7, 7 | 60.3 (9.01) | 62.9 (6.82)
  Part A, SA, Dose 1, 30 min, n=7, 7 | 59.1 (8.45) | 62.4 (7.16)
  Part A, SA, Dose 1, 1 hr, n=7, 7 | 62.6 (8.81) | 62.4 (6.35)
  Part A, SA, Dose 2 avg Pre-dose, n=7, 7 | 69.0 (7.84) | 70.6 (6.20)
  Part A, SA, Dose 2, 5 min, n=7, 7 | 66.7 (9.16) | 71.1 (8.19)
  Part A, SA, Dose 2, 15 min, n=7, 7 | 66.0 (7.37) | 69.6 (10.05)
  Part A, SA, Dose 2, 30 min, n=7, 7 | 65.1 (7.78) | 65.7 (6.99)
  Part A, SA, Dose 2, 1hr, n=7, 7 | 65.7 (7.06) | 68.6 (8.30)
  Part B, avg Pre-dose, n=10, 11 | 64.5 (6.21) | 68.4 (8.85)
  Part B, 5 min, n=10, 11 | 60.0 (6.18) | 65.9 (8.87)
  Part B, 15 min, n=10, 11 | 59.4 (4.99) | 63.5 (6.52)
  Part B, 1 hr, n=10, 11 | 58.6 (6.20) | 61.0 (6.07)
  Part C, avg Pre-dose, n=9, 9 | 62.4 (4.27) | 66.3 (7.07)
  Part C, 5 min, n=9, 9 | 60.3 (9.31) | 65.0 (9.15)
  Part C, 15 min, n=9, 9 | 60.8 (6.51) | 60.7 (5.50)
  Part C, 1hr, n=9, 9 | 59.2 (6.50) | 61.1 (6.47)

6. Secondary Outcome: Mean Body Temperature at the Indicated Time Points in Parts A, B and C
Description: Body temperature measurements were obtained at1 hr post-dose 2 FA and SA in Part A and each administration in Parts B, and C. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A.
Time Frame: 1 hr post the second dose administered in Part A and 1 hr post each dose administered in Parts B and C (up to 8 Weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
Degree Celsius
  Part A, FA, Dose 2, 1 hr, n=15, 12 | 36.84 (0.470) | 36.70 (0.484)
  Part A, SA, Dose 2, 1 hr, n=7, 7 | 36.56 (0.541) | 36.80 (0.520)
  Part B, 1 hr, n=10, 10 | 36.55 (0.536) | 36.76 (0.414)
  Part C, 1 hr, n=9, 9 | 36.54 (0.391) | 36.69 (0.473)

7. Secondary Outcome: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) Findings in Parts A, B and C
Description: A 12-lead ECG was recorded in a seated position after the participant was kept at rest in this position for at least 10 minutes. ECGs were obtained at pre-dose and 5 min, 15 min (only in Part A) 30 min, and 1 hr after FA and SA in Part A and each administration in Parts B, and C. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. Data are presented as clinically significant (CS) or not clinically significant (NCS) abnormal findings any time during study. The study investigator determined if the abnormal ECG finding was CS or NCS.
Time Frame: Pre-dose and 5min to 1 hr after each dose administered in Parts A, B and C (up to 8 Weeks)
Population: All subject population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
Participants
  Part A, FA, Normal, n=16, 14 | 13 | 12
  Part A, FA, Abnormal NCS, n=16, 14 | 2 | 2
  Part A, FA Abnormal CS, n=16, 14 | 1 | 0
  Part A, SA, Normal, n=7, 7 | 4 | 7
  Part A, SA, Abnormal NCS, n=7, 7 | 2 | 0
  Part A, SA, Abnormal CS, n=7, 7 | 1 | 0
  Part B, Normal, n=10, 11 | 9 | 10
  Part B, Abnormal NCS, n=10, 11 | 1 | 1
  Part B, Abnormal CS, n=10, 11 | 0 | 0
  Part C, Normal, n=9, 9 | 9 | 8
  Part C, Abnormal NCS, n=9, 9 | 0 | 1
  Part C, Abnormal CS, n=9, 9 | 0 | 0

8. Secondary Outcome: Mean Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count, and White Blood Cells (WBC) Count Values at the Indicated Time Points in Part A
Description: Blood samples were collected for the measurement of basophils, eosinophils, lymphocytes, monocytes, total neutrophils (ANC - absolute neutrophil count), platelet count, and white blood cells count at pre-dose and 1 hr after each dose of FA and SA in Part A. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A.
Time Frame: Pre-dose and 1 hr post each dose administered in Part A (up to 3 Weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^9 cells/Liter (GI/L)
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
10^9 cells/Liter (GI/L)
  Basophils, FA, Pre-dose, n=16, 14 | 0.026 (0.0126) | 0.023 (0.0159)
  Basophils, FA, 1 hr Post-dose, n=14, 13 | 0.031 (0.0192) | 0.032 (0.0242)
  Basophils, SA, Pre-dose, n=6, 7 | 0.040 (0.0329) | 0.026 (0.0162)
  Basophils, SA, 1 hr Post-dose, n=7, 7 | 0.019 (0.0107) | 0.036 (0.0299)
  Eosinophils, FA, Pre-dose, n=16, 14 | 0.091 (0.0604) | 0.063 (0.0365)
  Eosinophils, FA, 1 hr Post-dose, n=14, 13 | 0.106 (0.0776) | 0.093 (0.0471)
  Eosinophils, SA, Pre-dose, n=6, 7 | 0.080 (0.0510) | 0.064 (0.0299)
  Eosinophils, SA, 1 hr Post-dose, n=7, 7 | 0.113 (0.0502) | 0.080 (0.0191)
  Lymphocytes, FA, Pre-dose, n=16, 14 | 1.801 (0.4214) | 1.673 (0.3348)
  Lymphocytes, FA, 1 hr Post-dose, n=14, 13 | 2.095 (0.4572) | 1.977 (0.5392)
  Lymphocytes, SA, Pre-dose, n=6, 7 | 1.922 (0.4492) | 1.536 (0.3406)
  Lymphocytes, SA, 1 hr Post-dose, n=7, 7 | 2.200 (0.6387) | 1.926 (0.2486)
  Monocytes, FA, Pre-dose, n=16, 14 | 0.363 (0.1373) | 0.369 (0.1957)
  Monocytes, FA, 1 hr Post-dose, n=14, 13 | 0.414 (0.1249) | 0.434 (0.1601)
  Monocytes, SA, Pre-dose, n=6, 7 | 0.390 (0.1517) | 0.297 (0.0525)
  Monocytes, SA, 1 hr Post-dose, n=7, 7 | 0.380 (0.1319) | 0.364 (0.0479)
  Total Neutrophils, FA, Pre-dose, n=16, 14 | 4.256 (1.3244) | 4.206 (1.1230)
  Total Neutrophils, FA, 1 hr Post-dose, n=14, 13 | 4.730 (1.3512) | 4.800 (1.1399)
  Total Neutrophils, SA, Pre-dose, n=6, 7 | 4.238 (1.4993) | 3.993 (0.9757)
  Total Neutrophils, SA, 1 hr Post-dose, n=7, 7 | 4.847 (1.4473) | 4.250 (0.6064)
  Platelet count, FA, Pre-dose, n=16, 13 | 225.8 (51.14) | 233.4 (56.53)
  Platelet count, FA, 1 hr Post-dose, n=14, 13 | 209.1 (49.01) | 215.7 (30.69)
  Platelet count, SA, Pre-dose, n=6, 7 | 259.8 (36.98) | 238.6 (47.90)
  Platelet count, SA, 1 hr Post-dose, n=7, 7 | 238.4 (53.37) | 232.3 (49.45)
  WBC count, FA, Pre-dose, n=16, 14 | 6.54 (1.565) | 6.33 (1.315)
  WBC count, FA, 1 hr Post-dose, n=14, 13 | 7.36 (1.663) | 7.33 (1.596)
  WBC count, SA, Pre-dose, n=6, 7 | 6.67 (1.560) | 5.91 (1.263)
  WBC count, SA, 1 hr Post-dose, n=7, 7 | 7.53 (1.798) | 6.66 (0.810)

9. Secondary Outcome: Mean Hemoglobin, Mean Corpuscle Hemoglobin Concentration (MCHC), Albumin and Total Protein Values at the Indicated Time Points in Part A
Description: Blood samples were collected for the measurement of hemoglobin, MCHC, albumin and total protein at pre-dose and 1 hr after each dose of FA and SA in Part A. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A.
Time Frame: Pre-dose and 1 hr post each dose administered in Part A (up to 3 Weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Grams per liter (G/L)
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
Grams per liter (G/L)
  Hemoglobin, FA, Pre-dose, n=16, 14 | 134.1 (11.16) | 134.2 (11.82)
  Hemoglobin, FA, 1 hr Post-dose, n=14, 13 | 130.1 (11.35) | 130.5 (11.17)
  Hemoglobin, SA, Pre-dose, n=6, 7 | 127.5 (8.69) | 133.4 (10.34)
  Hemoglobin, SA, 1 hr Post-dose, n=7, 7 | 125.4 (9.64) | 129.6 (9.78)
  MCHC, FA, Pre-dose, n=16, 14 | 325.6 (5.76) | 326.3 (6.14)
  MCHC, FA, 1 hr Post-dose, n=14, 13 | 327.0 (4.91) | 329.2 (5.36)
  MCHC, SA, Pre-dose, n=6, 7 | 327.5 (7.20) | 324.0 (6.51)
  MCHC, SA, 1 hr Post-dose, n=7, 7 | 327.7 (5.09) | 323.3 (10.24)
  Albumin, FA, Pre-dose, n=16, 14 | 43.4 (3.10) | 43.1 (2.11)
  Albumin, FA, 1 hr Post-dose, n=14, 14 | 41.7 (2.23) | 41.6 (1.82)
  Albumin, SA, Pre-dose, n=6, 7 | 43.3 (3.27) | 43.6 (2.15)
  Albumin, SA, 1 hr Post-dose, n=7, 7 | 41.4 (2.30) | 41.6 (1.99)
  Total protein, FA, Pre-dose, n=16, 14 | 69.3 (4.32) | 68.5 (2.41)
  Total protein, FA, 1 hr Post-dose, n=14, 14 | 66.1 (3.35) | 66.6 (2.41)
  Total protein, SA, Pre-dose, n=6, 7 | 69.0 (4.69) | 69.1 (3.34)
  Total protein, SA, 1 hr Post-dose, n=7, 7 | 65.4 (4.16) | 66.0 (3.61)

10. Secondary Outcome: Mean Hematocrit Values at the Indicated Time Points in Part A
Description: Blood samples were collected for the measurement of hematocrit at pre-dose and 1 hr after each dose of FA and SA in Part A. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A.
Time Frame: Pre-dose and 1 hr post each dose administered in Part A (up to 3 Weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Proportion of one
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
Proportion of one
  FA, Pre-dose, n=16, 14 | 0.4126 (0.03824) | 0.4119 (0.04143)
  FA, 1 hr Post-dose, n=14, 13 | 0.3979 (0.03595) | 0.3973 (0.03701)
  SA, Pre-dose, n=6, 7 | 0.3895 (0.02894) | 0.4120 (0.03950)
  SA, 1 hr Post-dose, n=7, 7 | 0.3826 (0.03321) | 0.4010 (0.03316)

11. Secondary Outcome: Mean Corpuscle Hemoglobin Values at the Indicated Time Points in Part A
Description: Blood samples were collected for the measurement of mean corpuscle hemoglobin at pre-dose and 1 hr after each dose of FA and SA in Part A. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A.
Time Frame: Pre-dose and 1 hr post each dose administered in Part A (up to 3 Weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: picograms per cell (pg)
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
picograms per cell (pg)
  FA, Pre-dose, n=16, 14 | 29.87 (1.709) | 29.75 (1.787)
  FA, 1 hr Post-dose, n=14, 13 | 29.75 (1.874) | 29.85 (1.859)
  SA, Pre-dose, n=6, 7 | 29.48 (1.958) | 29.67 (1.627)
  SA, 1 hr Post-dose, n=7, 7 | 29.67 (1.864) | 29.40 (1.672)

12. Secondary Outcome: Mean Corpuscle Volume Values at the Indicated Time Points in Part A
Description: Blood samples were collected for the measurement of mean corpuscle volume at pre-dose and 1 hr after each dose of FA and SA in Part A. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A
Time Frame: Pre-dose and 1 hr post each dose administered in Part A (up to 3 Weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: femtoliters per cell (fL)
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
femtoliters per cell (fL)
  FA, Pre-dose, n=16, 14 | 91.8 (5.03) | 91.3 (5.21)
  FA, 1 hr Post-dose, n=14, 13 | 91.0 (5.04) | 90.8 (5.63)
  SA, Pre-dose, n=6, 7 | 90.0 (6.19) | 91.6 (5.49)
  SA, 1 hr Post-dose, n=7, 7 | 90.4 (5.72) | 91.2 (5.66)

13. Secondary Outcome: Mean Red Blood Cell Count Values at the Indicated Time Points in Part A
Description: Blood samples were collected for the measurement of red blood cell count at pre-dose and 1 hr after each dose of FA and SA in Part A. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A.
Time Frame: Pre-dose and 1 hr post each dose administered in Part A (up to 3 Weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (TI/L)
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
10^12 cells per liter (TI/L)
  FA, Pre-dose, n=16, 14 | 4.52 (0.452) | 4.54 (0.553)
  FA, 1 hr Post-dose, n=14, 13 | 4.40 (0.470) | 4.39 (0.460)
  SA, Pre-dose, n=6, 7 | 4.34 (0.296) | 4.51 (0.522)
  SA, 1 hr Post-dose, n=7, 7 | 4.24 (0.436) | 4.42 (0.406)

14. Secondary Outcome: Mean Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and Gamma Glutamyl Transferase (GGT) Values at the Indicated Time Points in Part A
Description: Blood samples were collected for the measurement of ALP, ALT, AST and GGT at pre-dose and 1 hr after each dose of FA and SA in Part A. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A.
Time Frame: Pre-dose and 1 hr post each dose administered in Part A (up to 3 Weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: International Units/Liter (IU/L)
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
International Units/Liter (IU/L)
  ALP, FA, Pre-dose, n=16, 14 | 67.9 (19.33) | 64.1 (15.01)
  ALP, FA, 1 hr Post-dose, n=14, 14 | 63.7 (16.70) | 60.6 (13.67)
  ALP, SA, Pre-dose, n=6, 7 | 69.7 (15.11) | 57.4 (13.36)
  ALP, SA, 1 hr Post-dose, n=7, 7 | 69.0 (17.45) | 55.9 (13.59)
  ALT, FA, Pre-dose, n=16, 14 | 15.8 (5.36) | 13.9 (4.62)
  ALT, FA, 1 hr Post-dose, n=14, 14 | 15.2 (5.83) | 14.1 (5.77)
  ALT, SA, Pre-dose, n=6, 7 | 16.5 (2.07) | 13.6 (5.74)
  ALT, SA, 1 hr Post-dose, n=7, 7 | 15.3 (2.75) | 12.9 (6.54)
  AST, FA, Pre-dose, n=16, 14 | 23.1 (10.37) | 19.6 (3.98)
  AST, FA, 1 hr Post-dose, n=14, 13 | 21.4 (9.87) | 20.7 (7.51)
  AST, SA, Pre-dose, n=6, 7 | 18.5 (4.28) | 21.6 (6.45)
  AST, SA, 1 hr Post-dose, n=6, 7 | 16.5 (3.51) | 19.7 (7.11)
  GGT, FA, Pre-dose, n=16, 14 | 24.6 (12.93) | 22.8 (9.95)
  GGT, FA, 1 hr Post-dose, n=14, 14 | 24.6 (13.89) | 22.4 (9.85)
  GGT, SA, Pre-dose, n=6, 7 | 20.7 (9.18) | 22.9 (12.82)
  GGT, SA, 1 hr Post-dose, n=7, 7 | 25.0 (15.58) | 22.0 (13.17)

15. Secondary Outcome: Mean Direct Bilirubin, Total Bilirubin, Creatinine and Uric Acid Values at the Indicated Time Points in Part A
Description: Blood samples were collected for the measurement ofdirect bilirubin, total bilirubin, creatinine and uric acid at pre-dose and 1 hr after each dose of FA and SA in Part A. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A.
Time Frame: Pre-dose and 1 hr post each dose administered in Part A (up to 3 Weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
Micromoles per liter (µmol/L)
  Direct bilirubin, FA, Pre-dose, n=13, 11 | 1.77 (0.832) | 1.64 (0.809)
  Direct bilirubin, FA, 1 hr Post-dose, n=10, 11 | 1.80 (0.919) | 1.45 (0.522)
  Direct bilirubin, SA, Pre-dose, n=4, 6 | 1.75 (0.957) | 1.83 (0.753)
  Direct bilirubin, SA, 1 hr Post-dose, n=5, 6 | 1.20 (0.447) | 1.50 (0.548)
  Total bilirubin, FA, Pre-dose, n=16, 14 | 8.07 (3.999) | 8.04 (3.709)
  Total bilirubin, FA, 1 hr Post-dose, n=14, 14 | 7.04 (4.185) | 6.34 (2.453)
  Total bilirubin, SA, Pre-dose, n=6, 7 | 7.35 (3.075) | 7.71 (2.928)
  Total bilirubin, SA, 1 hr Post-dose, n=7, 7 | 6.59 (3.204) | 5.87 (1.928)
  Creatinine, FA, Pre-dose, n=16, 14 | 65.1 (12.99) | 64.0 (11.21)
  Creatinine, FA, 1 hr Post-dose, n=14, 14 | 65.0 (12.29) | 60.5 (8.49)
  Creatinine, SA, Pre-dose, n=6, 7 | 61.1 (11.82) | 66.5 (11.72)
  Creatinine, SA, 1 hr Post-dose, n=7, 7 | 63.0 (10.92) | 65.1 (7.83)
  Uric acid, FA, Pre-dose, n=16, 14 | 283.1 (66.30) | 272.8 (59.36)
  Uric acid, FA, 1 hr Post-dose, n=14, 14 | 269.3 (68.09) | 259.2 (57.65)
  Uric acid, SA, Pre-dose, n=6, 7 | 270.0 (30.61) | 273.7 (74.40)
  Uric acid, SA, 1 hr Post-dose, n=7, 7 | 275.4 (43.08) | 257.7 (65.80)

16. Secondary Outcome: Mean Calcium, Chloride, Glucose, Potassium, Sodium, and Urea/Blood Urea Nitrogen (BUN) Values at the Indicated Time Points in Part A
Description: Blood samples were collected for the measurement of calcium, chloride, glucose, potassium, sodium, and urea/blood urea nitrogen (BUN) at pre-dose and 1 hr after each dose of FA and SA in Part A. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A.
Time Frame: Pre-dose and 1 hr post each dose administered in Part A (up to 3 Weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
Millimoles per liter (mmol/L)
  Calcium, FA, Pre-dose, n=16, 14 | 2.37 (0.085) | 2.39 (0.107)
  Calcium, FA, 1 hr Post-dose, n=14, 13 | 2.34 (0.099) | 2.34 (0.091)
  Calcium, SA, Pre-dose, n=6, 7 | 2.41 (0.102) | 2.37 (0.095)
  Calcium, SA, 1 hr Post-dose, n=6, 7 | 2.34 (0.061) | 2.32 (0.110)
  Chloride, FA, Pre-dose, n=16, 14 | 103.6 (2.31) | 103.4 (2.13)
  Chloride, FA, 1 hr Post-dose, n=14, 14 | 103.6 (2.06) | 104.3 (2.20)
  Chloride, SA, Pre-dose, n=6, 7 | 103.6 (3.02) | 103.0 (1.73)
  Chloride, SA, 1 hr Post-dose, n=7, 7 | 104.9 (4.26) | 103.6 (1.40)
  Glucose, FA, Pre-dose, n=16, 14 | 5.28 (0.884) | 5.19 (0.791)
  Glucose, FA, 1 hr Post-dose, n=14, 14 | 5.59 (1.124) | 5.69 (1.279)
  Glucose, SA, Pre-dose, n=6, 7 | 5.03 (1.108) | 5.06 (0.629)
  Glucose, SA, 1 hr Post-dose, n=7, 7 | 5.46 (1.165) | 5.24 (0.873)
  Potassium, FA, Pre-dose, n=16, 14 | 4.18 (0.246) | 4.18 (0.229)
  Potassium, FA, 1 hr Post-dose, n=14, 13 | 3.94 (0.318) | 4.55 (1.028)
  Potassium, SA, Pre-dose, n=6, 7 | 4.22 (0.240) | 4.11 (0.241)
  Potassium, SA, 1 hr Post-dose, n=6, 7 | 4.12 (0.736) | 3.93 (0.206)
  Sodium, FA, Pre-dose, n=16, 14 | 138.6 (1.59) | 138.9 (1.51)
  Sodium, FA, 1 hr Post-dose, n=14, 14 | 138.8 (1.93) | 138.1 (1.99)
  Sodium, SA, Pre-dose, n=6, 7 | 139.0 (1.26) | 138.4 (0.98)
  Sodium, SA, 1 hr Post-dose, n=7, 7 | 140.0 (4.58) | 138.7 (1.60)
  Urea/BUN, FA, Pre-dose, n=16, 14 | 4.91 (1.909) | 4.86 (1.934)
  Urea/BUN, FA, 1 hr Post-dose, n=14, 14 | 5.04 (2.008) | 5.21 (2.104)
  Urea/BUN, SA, Pre-dose, n=6, 7 | 4.03 (1.791) | 4.81 (1.732)
  Urea/BUN, SA, 1 hr Post-dose, n=7, 7 | 5.00 (2.309) | 5.24 (1.706)

17. Secondary Outcome: Mean Troponin I Values at the Indicated Time Points in Part A
Description: Blood samples were collected for the measurement of troponin I at pre-dose and 1 hr after each dose of FA and SA in Part A. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. Cardiac troponin values that were below the quantification limit [0.02 or 0.04 microgram (mcg/L)] were imputed as 0.01 (mcg/L).
Time Frame: Pre-dose and 1 hr post each dose administered in Part A (up to 3 Weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
mcg/L
  FA, Pre-dose, n=16, 14 | 0.011 (0.0034) | 0.010 (0.0000)
  FA, 1 hr Post-dose, n=15, 13 | 0.010 (0.0000) | 0.010 (0.0000)
  SA, Pre-dose, n=7, 7 | 0.010 (0.0000) | 0.010 (0.0000)
  SA, 1 hr Post-dose, n=7, 7 | 0.010 (0.0000) | 0.010 (0.0000)

18. Secondary Outcome: Mean Forced Expiratory Volume in One Second (FEV1) Values at the Indicated Time Points in Parts A, B and C
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. FEV1 was measured by spirometry at pre-dose and 30 min after FA and SA in Part A and each administration in Parts B, and C. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A.
Time Frame: Pre-dose and 30 min post each dose administered in Parts A, B and C (up to 8 Weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
Liters
  Part A, FA, Dose 1, Pre-dose, n=16, 14 | 2.55 (2.18) | 2.43 (2.17)
  Part A, FA, Dose 1, 30 min Post-dose, n=16, 14 | 2.49 (2.12) | 2.39 (2.10)
  Part A, FA, Dose 2, Pre-dose, n=16, 14 | 2.55 (2.22) | 2.37 (2.10)
  Part A, FA, Dose 2, 30 min Post-dose, n=15, 13 | 2.44 (2.06) | 2.29 (2.02)
  Part A, SA, Dose 1, Pre-dose, n=7, 7 | 2.54 (2.16) | 2.44 (1.97)
  Part A, SA, Dose 1, 30 min Post-dose, n=7, 7 | 2.42 (2.00) | 2.31 (1.76)
  Part A, SA, Dose 2, Pre-dose, n=7, 7 | 2.41 (1.99) | 2.36 (1.83)
  Part A, SA, Dose 2, 30 min Post-dose, n=7, 7 | 2.42 (1.97) | 2.32 (1.80)
  Part B, Pre-dose, n=10, 11 | 2.26 (2.07) | 2.31 (2.05)
  Part B, 30 min Post-dose, n=10, 11 | 2.17 (2.01) | 2.30 (2.05)
  Part C, Pre-dose, n=9, 9 | 2.23 (2.08) | 2.24 (1.98)
  Part C, 30 min Post-dose, n=9, 9 | 2.13 (1.96) | 2.22 (1.98)

19. Secondary Outcome: Number of Participants With Perception of Change in Oropharyngeal Sensation at the Indicated Time Points in Part A
Description: The perception of change in oropharyngeal sensation was assessed by a 4 point scale where participants were asked to describe sensitivity and perception of numbness and the responses were recorded. The following information was collected: 0 = no anaesthesia (A), 1 = mild anaesthesia, 2 = moderate anaesthesia and 3 = severe anaesthesia. Oropharyngeal examination was performed at 2 min, 5 min, 15 min, 30 min, 1 hr and 2 hr after FA and SA in Part A. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A
Time Frame: From 2 min -2 hr post each dose administered at Visits 1, 2 and 3 in Part A (up to 8 weeks)
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
Participants
  No A, FA, Dose 1, 2 min Post-dose, n=16, 14 | 16 | 14
  No A, FA, Dose 1, 5 min Post-dose, n=16, 14 | 16 | 14
  No A, FA, Dose 1, 15 min Post-dose, n=16, 14 | 16 | 14
  No A, FA, Dose 1, 30 min Post-dose, n=16, 14 | 16 | 14
  No A, FA, Dose 1, 1 hr Post-dose, n=16, 14 | 16 | 14
  No A, FA, Dose 2, 2 min Post-dose, n=15, 14 | 15 | 14
  No A, FA, Dose 2, 5 min Post-dose, n=15, 14 | 15 | 14
  No A, FA, Dose 2, 15 min Post-dose, n=15, 14 | 15 | 14
  No A, FA, Dose 2, 30 min Post-dose, n=15, 14 | 15 | 14
  No A, FA, Dose 2, 1 hr Post-dose, n=15, 14 | 15 | 14
  No A, SA, Dose 1, 2 min Post-dose, n=7, 7 | 7 | 7
  No A, SA, Dose 1, 5 min Post-dose, n=7, 7 | 7 | 7
  No A, SA, Dose 1, 15 min Post-dose, n=7, 7 | 7 | 7
  No A, SA, Dose 1, 30 min Post-dose, n=7, 7 | 7 | 7
  No A, SA, Dose 1, 1 hr Post-dose, n=7,7 | 7 | 7
  No A, SA, Dose 2, 2 min Post-dose, n=7, 7 | 7 | 7
  No A, SA, Dose 2, 5 min Post-dose, n=7, 7 | 7 | 7
  No A, SA, Dose 2, 15 min Post-dose, n=7, 7 | 7 | 7
  No A, SA, Dose 2, 30 min Post-dose, n=7, 7 | 7 | 7
  No A, SA, Dose 2, 1 hr Post-dose, n=7, 7 | 7 | 7
  Mild A, FA, Dose 1, 2 min Post-dose, n=16, 14 | 0 | 0
  Mild A, FA, Dose 1, 5 min Post-dose, n=16, 14 | 0 | 0
  Mild A, FA, Dose 1, 15 min Post-dose, n=16, 14 | 0 | 0
  Mild A, FA, Dose 1, 30 min Post-dose, n=16, 14 | 0 | 0
  Mild A, FA, Dose 1, 1 hr Post-dose, n=16, 14 | 0 | 0
  Mild A, FA, Dose 2, 2 min Post-dose, n=15, 14 | 0 | 0
  Mild A, FA, Dose 2, 5 min Post-dose, n=15, 14 | 0 | 0
  Mild A, FA, Dose 2, 15 min Post-dose, n=15, 14 | 0 | 0
  Mild A, FA, Dose 2, 30 min Post-dose, n=15, 14 | 0 | 0
  Mild A, FA, Dose 2, 1 hr Post-dose, n=15, 14 | 0 | 0
  Mild A, SA, Dose 1, 2 min Post-dose, n=7, 7 | 0 | 0
  Mild A, SA, Dose 1, 5 min Post-dose, n=7, 7 | 0 | 0
  Mild A, SA, Dose 1, 15 min Post-dose, n=7, 7 | 0 | 0
  Mild A, SA, Dose 1, 30 min Post-dose, n=7, 7 | 0 | 0
  Mild A, SA, Dose 1, 1 hr Post-dose, n=7,7 | 0 | 0
  Mild A, SA, Dose 2, 2 min Post-dose, n=7, 7 | 0 | 0
  Mild A, SA, Dose 2, 5 min Post-dose, n=7, 7 | 0 | 0
  Mild A, SA, Dose 2, 15 min Post-dose, n=7, 7 | 0 | 0
  Mild A, SA, Dose 2, 30 min Post-dose, n=7, 7 | 0 | 0
  Mild A, SA, Dose 2, 1 hr Post-dose, n=7, 7 | 0 | 0
  Moderate A, FA, Dose 1, 2 min Post-dose, n=16, 14 | 0 | 0
  Moderate A, FA, Dose 1, 5 min Post-dose, n=16, 14 | 0 | 0
  Moderate A, FA, Dose 1, 15 min Post-dose, n=16, 14 | 0 | 0
  Moderate A, FA, Dose 1, 30 min Post-dose, n=16, 14 | 0 | 0
  Moderate A, FA, Dose 1, 1 hr Post-dose, n=16, 14 | 0 | 0
  Moderate A, FA, Dose 2, 2 min Post-dose, n=15, 14 | 0 | 0
  Moderate A, FA, Dose 2, 5 min Post-dose, n=15, 14 | 0 | 0
  Moderate A, FA, Dose 2, 15 min Post-dose, n=15, 14 | 0 | 0
  Moderate A, FA, Dose 2, 30 min Post-dose, n=15, 14 | 0 | 0
  Moderate A, FA, Dose 2, 1 hr Post-dose, n=15, 14 | 0 | 0
  Moderate A, SA, Dose 1, 2 min Post-dose, n=7, 7 | 0 | 0
  Moderate A, SA, Dose 1, 5 min Post-dose, n=7, 7 | 0 | 0
  Moderate A, SA, Dose 1, 15 min Post-dose, n=7, 7 | 0 | 0
  Moderate A, SA, Dose 1, 30 min Post-dose, n=7, 7 | 0 | 0
  Moderate A, SA, Dose 1, 1 hr Post-dose, n=7,7 | 0 | 0
  Moderate A, SA, Dose 2, 2 min Post-dose, n=7, 7 | 0 | 0
  Moderate A, SA, Dose 2, 5 min Post-dose, n=7, 7 | 0 | 0
  Moderate A, SA, Dose 2, 15 min Post-dose, n=7, 7 | 0 | 0
  Moderate A, SA, Dose 2, 30 min Post-dose, n=7, 7 | 0 | 0
  Moderate A, SA, Dose 2, 1 hr Post-dose, n=7, 7 | 0 | 0
  Severe A, FA, Dose 1, 2 min Post-dose, n=16, 14 | 0 | 0
  Severe A, FA, Dose 1, 5 min Post-dose, n=16, 14 | 0 | 0
  Severe A, FA, Dose 1, 15 min Post-dose, n=16, 14 | 0 | 0
  Severe A, FA, Dose 1, 30 min Post-dose, n=16, 14 | 0 | 0
  Severe A, FA, Dose 1, 1 hr Post-dose, n=16, 14 | 0 | 0
  Severe A, FA, Dose 2, 2 min Post-dose, n=15, 14 | 0 | 0
  Severe A, FA, Dose 2, 5 min Post-dose, n=15, 14 | 0 | 0
  Severe A, FA, Dose 2, 15 min Post-dose, n=15, 14 | 0 | 0
  Severe A, FA, Dose 2, 30 min Post-dose, n=15, 14 | 0 | 0
  Severe A, FA, Dose 2, 1 hr Post-dose, n=15, 14 | 0 | 0
  Severe A, SA, Dose 1, 2 min Post-dose, n=7, 7 | 0 | 0
  Severe A, SA, Dose 1, 5 min Post-dose, n=7, 7 | 0 | 0
  Severe A, SA, Dose 1, 15 min Post-dose, n=7, 7 | 0 | 0
  Severe A, SA, Dose 1, 30 min Post-dose, n=7, 7 | 0 | 0
  Severe A, SA, Dose 1, 1 hr Post-dose, n=7, 7 | 0 | 0
  Severe A, SA, Dose 2, 2 min Post-dose, n=7, 7 | 0 | 0
  Severe A, SA, Dose 2, 5 min Post-dose, n=7, 7 | 0 | 0
  Severe A, SA, Dose 2, 15 min Post-dose, n=7, 7 | 0 | 0
  Severe A, SA, Dose 2, 30 min Post-dose, n=7, 7 | 0 | 0
  Severe A, SA, Dose 2, 1 hr Post-dose, n=7, 7 | 0 | 0

20. Secondary Outcome: Mean Transient Cough Counts at the Indicated Time Points in Part A
Description: Cough counts (8 hours of recording) was conducted at Visits 1, 2 and 3 (4 hours of post-dose recording for each of the two doses administered). Coughs was counted by a cough monitor fitted to the participants for 8 hours post Dose 1. Transient coughing was calculated as the total number of coughs experienced in the two minutes from the start of the first inhalation of a dose. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A
Time Frame: 0-4 hr, 4-8 hr, 0-8 hr post each dose at Visits 1, 2 and 3 in Part A (up to 8 weeks)
Population: All Subjects Population.Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed for different time points, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: Cough count
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 14 | 14
Cough count
  FA, 0-4 hr, n=14, 14 | 1.7 (3.41) | 17.8 (16.27)
  FA, 4-8 hr, n=14, 14 | 0.9 (1.88) | 19.0 (10.91)
  FA, 0-8 hr, n=14, 14 | 2.6 (4.11) | 36.8 (25.41)
  SA, 0-4 hr, n=7, 7 | 0.0 (0.0) | 18.3 (13.51)
  SA, 4-8 hr, n=7, 7 | 2.0 (3.42) | 15.9 (12.02)
  SA, 0-8 hr, n=7, 7 | 2.0 (3.42) | 34.1 (24.83)

21. Secondary Outcome: Plasma Concentrations of GSK2339345 at the Indicated Time Points at Visits 1, 2 and 3 (Part A)
Description: Plasma concentrations of GSK2339345 following the first dose and second dose at each visit in Part A was measured. Samples were collected at the following time points: pre-dose, 2 min, 5 min, 10 min, 30 min, 1 hr and 2 hr (only after Dose 1) after each dose administration at Visits 1, 2 and 3. All non-quantifiable (NQ) values after the pre-first dose value imputed to half lower limit of quantification (LLQ) (LLQ=0.2 nanogram per milliliter [ng/mL]). Different participants may have been analyzed for different parameters, so the overall number of par. analyzed reflects everyone in the pharmacokinetic population.
Time Frame: From 0-4 hr post each dose administered at Visits 1, 2 and 3 in Part A (up to 3 weeks)
Population: The Pharmacokinetic (PK) Population comprised of participants in the All Subjects Population for whom a pharmacokinetic sample was obtained and analysed. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Median (Full Range); unit: nanogram per milliliter (ng/mL)
Arm/Group | GSK2339345 1000 µg
Number analyzed (Participants) | 14
nanogram per milliliter (ng/mL)
  FA, Dose 1, Pre-dose, n=14 | 0.000 [0.000 to 0.000]
  FA, Dose 1, 2 min Post-dose, n=14 | 1.3985 (1.4881) [0.100 to 5.540]
  FA, Dose 1, 5 min Post-dose, n=14 | 0.9565 (0.9955) [0.100 to 2.886]
  FA, Dose 1, 10 min Post-dose, n=14 | 0.6925 (0.5075) [0.100 to 1.522]
  FA, Dose 1, 30 min Post-dose, n=14 | 0.2820 (NA) [0.100 to 0.628]
  FA, Dose 1, 1 hr Post-dose, n=13 | 0.2950 (NA) [0.100 to 0.559]
  FA, Dose 1, 2 hr Post-dose, n=13 | 0.2010 (NA) [0.100 to 0.421]
  FA, Dose 2, 2 min Post-dose, n=14 | 1.8735 (3.4305) [0.100 to 13.483]
  FA, Dose 2, 5 min Post-dose, n=14 | 1.4315 (2.3894) [0.100 to 9.686]
  FA, Dose 2, 10 min Post-dose, n=14 | 1.0740 (0.9082) [0.100 to 3.119]
  FA, Dose 2, 30 min Post-dose, n=13 | 0.5230 (0.4645) [0.100 to 1.745]
  FA, Dose 2, Pre-dose, n=14 | 0.1000 [0.100 to 0.705]
  FA, Dose 2, 1 hr Post-dose, n=14 | 0.5475 (0.2788) [0.100 to 0.989]
  SA, Dose 1, Pre-dose, n=7 | 0.0000 (NA) [0.0000 to 0.441]
  SA, Dose 1, 2 min Post-dose, n=7 | 1.5010 (1.6036) [0.100 to 3.877]
  SA, Dose 1, 5 min Post-dose, n=7 | 1.5680 (1.0466) [0.100 to 2.642]
  SA, Dose 1, 10 min Post-dose, n=7 | 0.7790 (0.5366) [0.100 to 1.351]
  SA, Dose 1, 30 min Post-dose, n=7 | 0.2470 (3.1688) [0.100 to 8.619]
  SA, Dose 1, 1 hr Post-dose, n=7 | 0.2900 (0.1135) [0.100 to 0.380]
  SA, Dose 1, 2 hr Post-dose, n=7 | 0.1000 (NA) [0.100 to 0.826]
  SA, Dose 2, Pre-dose, n=7 | 0.1000 (NA) [0.100 to 0.541]
  SA, Dose 2, 2 min Post-dose, n=7 | 1.8280 (3.0811) [0.100 to 9.026]
  SA, Dose 2, 5 min Post-dose, n=7 | 1.4750 (1.7052) [0.100 to 5.130]
  SA, Dose 2, 10 min Post-dose, n=7 | 0.9030 (0.8469) [0.100 to 2.603]
  SA, Dose 2, 30 min Post-dose, n=7 | 0.4260 (NA) [0.100 to 0.737]
  SA, Dose 2, 1 hr Post-dose, n=7 | 0.4290 (0.4640) [0.100 to 1.456]

22. Secondary Outcome: Area Under the Concentration (AUC) Time (0-1) and AUC(0-t) of GSK2339345 Following Two Repeated Doses
Description: AUC curve from time zero (pre-dose) to 1 hours AUC(0-1) and from time zero to the last time AUC(0-t) of quantifiable concentration of GSK2339345 following the first dose and second dose at each visit in Part A was measured. Samples were collected at the following time points: pre-dose; 2 min, 5 min, 10 min, 30 min, 1 hr and 2hr (only after Dose 1) post every dose administration at Visits 1, 2 and 3. For , AUC(0-1) and AUC(0-t), non calculable (NC) were imputed prior to derivation of summary statistics and NCs were imputed as 0.1093 and 0.0855 respectively (=half the lowest observed value).
Time Frame: From 0-4 hr post each dose administered at Visits 1, 2 and 3 in Part A (up to 3 weeks)
Population: PK Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | GSK2339345 1000 µg
Number analyzed (Participants) | 14
hour*nanogram per milliliter (h*ng/mL)
  AUC(0-1), FA, Dose 1, n=11 | 0.3968 (109.1924)
  AUC(0-1), FA, Dose 2, n=10 | 0.8168 (76.8324)
  AUC(0-1), SA, Dose 1, n=7 | 0.4509 (174.9418)
  AUC(0-1), SA, Dose 2, n=6 | NA (NA) — Due to insufficient data, NA was entered.
  AUC(0-t), FA, n=14 | 2.0076 (174.1325)
  AUC(0-t), SA, n=7 | 1.2425 (559.1820)

23. Secondary Outcome: Maximum Observed Concentration (Cmax) of GSK2339345 Following Two Repeated Doses
Description: Cmax is defined as the maximum observed concentration of GSK2339345 following two repeated doses at each visit in Part A. Samples were collected at the following time points: pre-dose; 2 min, 5 min, 10 min, 30 min, 1 hr and 2hr (only after Dose 1) post every dose administration at Visits 1, 2 and 3. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. For Cmax, NCs were imputed prior to derivation of summary statistics and NCs were imputed with 0.5*LLQ (LLQ=0.20 ng/mL).
Time Frame: From 0-4 hr post each dose administered at Visits 1, 2 and 3 in Part A (up to 3 weeks)
Population: PK Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed for different time points, so the overall number of participants analyzed reflects everyone in the PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | GSK2339345 1000 µg
Number analyzed (Participants) | 14
nanogram per milliliter (ng/mL)
  FA, Dose 1, n=14 | 0.9485 (224.0451)
  FA, Dose 2, n=14 | 1.9212 (138.2018)
  SA, Dose 1, n=7 | 1.0835 (474.4072)
  SA, Dose 2, n=7 | 1.0448 (416.3398)

24. Secondary Outcome: Time to Reach the Observed Maximum Concentration (Tmax) of GSK2339345 Following Two Repeated Doses
Description: Tmax is defined as the time to reach the observed maximum GSK2339345concentration following two repeated doses at each visit in Part A. Samples were collected at the following time points: pre-dose; 2 min, 5 min, 10 min, 30 min, 1 hr and 2hr (only after Dose 1) post every dose administered at Visits 1, 2 and 3. FA is the first of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A. SA is the second of the two doses of GSK2339345 or placebo administered at any of the three visits in Part A.
Time Frame: From 0-4 hr post each dose administered at Visits 1, 2 and 3 in Part A (up to 3 weeks)
Population: as for outcome 23
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2339345 1000 µg
Number analyzed (Participants) | 14
Hours
  FA, Dose 1, n=11 | 0.03333 [0.0167 to 0.100]
  FA, Dose 2, n=14 | 0.03333 [0.0167 to 0.516]
  SA, Dose 1, n=5 | 0.06667 [0.0333 to 0.416]
  SA, Dose 2, n=5 | 0.03333 [0.0167 to 1.050]

25. Secondary Outcome: Mean Cough Count Over 4 Hours at Visits 1, 2 and 3 (Part A)
Description: Total cough count (8 hr of recording) was conducted at Visits 1, 2 and 3 (4- hrs of post-dose recording for each of the two doses administered). Coughs were counted by a cough monitor fitted to the participants for 8 hr post Dose 1. The cough count over 4-hrs was done by using the sum of first 4-hrs starting from the time of first dose and the second 4-hrs starting at the time of the second dose respectively. Number of coughs in 0-4 hr and 4-8 hr period was log-e transformed and used for the analysis. Values were imputed pro-rata if 4 hr epoch was less than 4 hr. Mean of the total cough counts over 4-hrs recorded post dose of every treatment i.e. placebo or GSK2339345 1000 mcg was reported.
Time Frame: Up to 8 hours post-dose at Visits 1, 2 and 3 (Part A)
Population: All Subjects Population. Only participants with at least one 4 hr cough count were analyzed.
Measure: Geometric Mean (Standard Error); unit: Cough count
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 14 | 14
Cough count
  0-4 hr | 70.5 (0.257) | 86.7 (0.257)
  4-8 hr | 65.1 (0.234) | 88.4 (0.234)
Statistical Analysis 1: Comparison: Placebo vs GSK2339345 1000 µg; Test type: Superiority or Other; Ratio of adjusted geometric mean = 1.23, 90% CI 2-sided [0.86 to 1.75] — Ratio of adjusted geometric means = GSK2339345/Placebo. Estimated value and CI are presented for the mean cough count over 0-4 hr
Statistical Analysis 2: Comparison: Placebo vs GSK2339345 1000 µg; Test type: Superiority or Other; Ratio of adjusted geometric mean = 1.36, 90% CI 2-sided [1.07 to 1.72] — Ratio of adjusted geometric means = GSK2339345/Placebo. Estimated value and CI are presented for the mean cough count over 4-8 hr

26. Secondary Outcome: Total Cough Count Excluding Transient Coughs Over 4 Hours at Visits 1, 2 and 3 (Part A)
Description: Total cough count (8 hr of recording) was conducted at Visits 1, 2 and 3 (4-hrs of post-dose recording for each of the two doses administered). Coughs were counted by a cough monitor fitted to the participants for 8 hr post Dose 1. Total count excluding transient cough over 4-hrs was done by using the sum of first 4-hrs starting from the time of first dose and the second 4-hrs starting at the time of the second dose respectively. Number of coughs excluding transient cough in 0-4 hr and 4-8 hr period was log-e transformed and used for the analysis. Values were imputed pro-rata if 4-hr epoch was less than 4-hrs. Mean of the total cough counts over 4-hrs recorded post dose of every treatment i.e. placebo or GSK2339345 1000 mcg was reported.
Time Frame: Up to 8 hours post-dose at Visits 1, 2 and 3 (Part A)
Population: All Subjects Population. Only participants with at least one 4 hr cough count were analyzed.
Measure: Geometric Mean (Standard Error); unit: Cough count
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 14 | 14
Cough count
  0-4 Hr | 70.2 (0.270) | 68.3 (0.270)
  4-8 Hr | 64.6 (0.250) | 67.0 (0.250)
Statistical Analysis 1: Comparison: Placebo vs GSK2339345 1000 µg; Test type: Superiority or Other; Ratio of adjusted geometric mean = 0.97, 90% CI 2-sided [0.67 to 1.40] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs GSK2339345 1000 µg; Test type: Superiority or Other; Ratio of adjusted geometric mean; Ratio of adjusted geometric means = GSK2 = 1.04, 90% CI 2-sided [0.79 to 1.36]

27. Secondary Outcome: Mean Cough Counts by 1 hr Epoch at Visits 1, 2 and 3 (Part A)
Description: Cough counts (8 hr of recording) were conducted at Visits 1, 2 and 3 (4-hr of post-dose recording for each of the two doses administered). Coughs were counted by a cough monitor fitted to the participant for 8 hr post Dose 1. The first epoch started at the time of the first dose, and the 60 min time periods continued until an epoch ended immediately before the second dose (or 4-hr after the first dose if earlier). The epochs were then re-started at the start of the second dose at 60 min intervals, finishing with an epoch which ran to 4-hrs after the start of the second dose. The cough counts were sum-up by the treatments received by the participants. Mean cough count was calculated per participant if the same treatment was taken during different periods. Values were imputed pro-rata if 1 hr epoch is less than 60 min.
Time Frame: Up to 8 hours post-dose at Visits 1, 2 and 3 in Part A (up to 3 weeks)
Population: All Subjects Population. Only those participants with a 1 hr cough count value were analyzed.
Measure: Mean (Standard Deviation); unit: Cough count
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 14 | 14
Cough count
  0 to 1 hr | 41.5 (30.25) | 46.8 (35.58)
  1 to 2 hr | 13.9 (9.86) | 15.7 (11.20)
  2 to 3 hr | 11.0 (11.68) | 17.0 (11.75)
  3 to 4 hr | 38.4 (35.63) | 36.6 (26.40)
  4 to 5 hr | 20.4 (14.78) | 54.7 (61.49)
  5 to 6 hr | 25.3 (43.09) | 28.9 (51.83)
  6 to 7 hr | 28.7 (44.03) | 18.7 (22.79)
  7 to 8 hr | 32.5 (54.26) | 28.2 (42.78)

28. Secondary Outcome: Mean Cough Counts by 30 Min Epoch at Visits 1, 2 and 3 (Part A)
Description: Cough counts (8 hr of recording) were conducted at Visits 1, 2 and 3 (4-hr of post-dose recording for each of the two doses administered). Coughs were counted by a cough monitor fitted to the participant for 8 hr post Dose 1. The first epoch started at the time of the first dose, and the 30 min time periods continued until an epoch ended immediately before the second dose (or 4-hr after the first dose if earlier). The epochs were then re-started at the start of the second dose at 30 min intervals, finishing with an epoch which ran to 4-hr after the start of the second dose. The cough counts were sum-up by the treatments received by the participants. Mean cough count was calculated per participant if the same treatment was taken during different periods.
Time Frame: Up to 8 hours post-dose in Visits 1, 2 and 3 in Part A (up to 3 weeks)
Population: All Subjects Population. Only those participants with a 30 min cough count value were analyzed.
Measure: Mean (Standard Deviation); unit: Cough count
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 14 | 14
Cough count
  0 to 0.5 hr | 15.3 (17.93) | 25.7 (21.17)
  0.5 to 1 hr | 26.2 (22.58) | 21.1 (22.18)
  1 to 1.5 hr | 7.1 (7.80) | 9.1 (8.29)
  1.5 to 2 hr | 6.7 (4.86) | 6.6 (6.10)
  2 to 2.5 hr | 5.9 (8.35) | 10.4 (10.29)
  2.5 to 3 hr | 5.1 (7.41) | 6.6 (8.67)
  3 to 3.5 hr | 19.2 (21.84) | 16.5 (15.60)
  3.5 to 4 hr | 19.2 (28.72) | 20.1 (23.39)
  4 to 4.5 hr | 5.4 (6.24) | 35.5 (44.15)
  4.5 to 5 hr | 15.0 (12.17) | 19.2 (21.38)
  5 to 5.5 hr | 19.1 (31.94) | 21.1 (49.66)
  5.5 to 6 hr | 6.2 (11.75) | 7.8 (10.60)
  6 to 6.5 hr | 12.0 (17.57) | 7.4 (8.26)
  6.5 to 7 hr | 16.7 (29.71) | 11.3 (16.92)
  7 to 7.5 hr | 16.5 (18.71) | 11.4 (15.10)
  7.5 to 8 hr | 16.0 (37.36) | 16.6 (33.54)

29. Secondary Outcome: Mean Cough Counts by 15 Min Epoch in Part A
Description: Cough counts (8 hr of recording) were conducted at Visits 1, 2 and 3 (4-hr of post-dose recording for each of the two doses administered). Coughs were counted by a cough monitor fitted to the participant for 8 hr post Dose 1. The first epoch started at the time of the first dose, and the 15 min time periods continued until an epoch ended immediately before the second dose (or 4h after the first dose if earlier). The epochs were then re-started at the start of the second dose at 15 min intervals, finishing with an epoch which ran to 4-hr after the start of the second dose. The cough counts were sum-up by the treatments received by the participants. Mean cough count was calculated per participant if the same treatment was taken during different periods.
Time Frame: Up to 8 hours post-dose at Visits 1, 2 and 3 in Part A (up to 3 weeks)
Population: All Subjects Population. Only those participants with a 15 min cough count value were analyzed.
Measure: Mean (Standard Deviation); unit: Cough count
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 14 | 14
Cough count
  0 to 0.25 hr | 4.6 (7.84) | 21.1 (18.23)
  0.25 to 0.5 hr | 10.7 (14.99) | 4.6 (9.21)
  0.5 to 0.75 hr | 22.5 (21.10) | 18.7 (19.54)
  0.75 to 1 hr | 3.7 (6.11) | 2.4 (3.91)
  1 to 1.25 hr | 4.9 (7.53) | 5.7 (6.91)
  1.25 to 1.5 hr | 2.3 (4.13) | 3.5 (4.19)
  1.5 to 1.75 hr | 3.5 (3.08) | 3.4 (3.67)
  1.75 to 2 hr | 3.3 (2.96) | 3.1 (3.61)
  2 to 2.25 hr | 4.0 (7.26) | 6.9 (9.04)
  2.25 to 2.5 hr | 1.9 (3.04) | 3.5 (4.77)
  2.5 to 2.75 hr | 0.4 (0.94) | 1.5 (4.39)
  2.75 to 3 hr | 4.6 (7.26) | 5.1 (6.34)
  3 to 3.25 hr | 8.4 (14.45) | 8.8 (13.61)
  3.25 to 3.5 hr | 10.9 (13.44) | 7.7 (11.34)
  3.5 to 3.75 hr | 7.7 (11.21) | 5.5 (8.60)
  3.75 to 4 hr | 11.5 (20.13) | 14.6 (21.35)
  4 to 4.25 hr | 1.6 (2.88) | 23.0 (17.97)
  4.25 to 4.5 hr | 3.8 (5.97) | 12.5 (28.66)
  4.5 to 4.75 hr | 12.4 (13.16) | 15.6 (19.11)
  4.75 to 5 hr | 2.6 (4.79) | 3.5 (5.51)
  5 to 5.25 hr | 9.6 (17.34) | 12.0 (28.61)
  5.25 to 5.5 hr | 9.5 (16.54) | 9.1 (21.65)
  5.5 to 5.75 hr | 2.1 (3.35) | 3.9 (6.34)
  5.75 to 6 hr | 4.1 (8.91) | 3.9 (6.24)
  6 to 6.25 hr | 6.8 (13.83) | 3.2 (4.39)
  6.25 to 6.5 hr | 5.2 (6.60) | 4.3 (6.01)
  6.5 to 6.75 hr | 7.2 (14.53) | 2.8 (4.67)
  6.75 to 7 hr | 9.5 (16.17) | 8.5 (12.80)
  7 to 7.25 hr | 6.9 (7.63) | 7.1 (11.20)
  7.25 to 7.5 hr | 9.6 (15.81) | 4.3 (5.51)
  7.5 to 7.75 hr | 6.9 (18.06) | 4.9 (6.24)
  7.75 to 8 hr | 9.1 (19.35) | 11.7 (33.10)

30. Secondary Outcome: Mean Visual Analogue Scale (VAS) Score of Cough Severity and Urge to Cough at the Indicated Time Points at Visits 1, 2 and 3 (Part A)
Description: VAS for urge to cough and severity of cough were recorded prior to first dose and 1 hour following the second dose of GSK2339345 or placebo at Visits 1, 2 and 3.VAS is a 100-mm linear scales on which participants indicated the severity of their cough (0 mm represents no severity and 100 mm maximum severity ever experienced) and urge to cough (0 represents no urge to cough, 100 represents maximum urge to cough ever experienced). Mean of replicate values per participants used where the same treatment taken during different periods.
Time Frame: Prior to first dose and 1hr post second dose at Visits 1, 2 and 3 in Part A (up to 3 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 16 | 14
Scores on a scale
  Urge to cough, Dose 1, Pre-dose, n=16, 14 | 42.9 (20.51) | 42.2 (25.94)
  Urge to cough, Dose 2, 1 hr Post-dose, n=15, 14 | 25.1 (15.40) | 41.5 (22.60)
  Cough severity, Dose 1, Pre-dose, n=16, 14 | 42.8 (16.71) | 37.3 (23.03)
  Cough severity, Dose 2, 1 hr Post-dose, n=15, 14 | 26.7 (15.03) | 39.3 (21.70)

31. Secondary Outcome: Mean Number of Cough Counts at Each Dose of the Challenge Agent for the Capsaicin Challenge (CC) at Visits 4 and 5 (Part B)
Description: Capsaicin was administered using a dosimeter through a nebulizer pot with flow-limitation. Inhalation of increased concentrations (Conc.) was continued until the maximum dose was tolerated by the par. or highest available Conc. was used. The dose-response relationship between dose of capsaicin and cough response was investigated using non-linear mixed effect modeling using Poisson and Negative Binomial distributions. When using a Poisson distribution, there was some evidence for a reduction in capsaicin Emax with GSK2339345 of 17.6%, however, this was not confirmed when using a Negative Binomial distribution. The Negative Binomial distribution described the data marginally better, but the dataset was too small to make definitive conclusions. There was no treatment difference in capsaicin ED50.
Time Frame: After the administration of GSK2339345 or placebo (first and second 15 seconds following each dose) at Visits 4 and 5 in Part B (up to 2 weeks)
Population: CC population. Population comprised of par. in the All Subjects Population for whom any CC data were available for one or both Part B study visits. Only those participants available at the specified time points we re analyze d (represented by n=X, X in the category titles).
Measure: Mean (Standard Deviation); unit: Cough count
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 10 | 11
Cough count
  0 to 15 sec, CC Conc.0.49 µmol/L, n=10, 11 | 0.0 (0.00) | 0.3 (0.90)
  0 to 15 sec, CC Conc.0.97 µmol/L, n=10, 11 | 0.0 (0.00) | 0.2 (0.60)
  0 to 15 sec, CC Conc.1.95 µmol/L, n=10, 11 | 2.0 (4.64) | 1.8 (3.19)
  0 to 15 sec, CC Conc.3.9 µmol/L, n=10, 11 | 4.7 (5.79) | 3.3 (6.20)
  0 to 15 sec, CC Conc. 7.81 µmol/L, n=10, 11 | 5.1 (6.45) | 5.3 (6.08)
  0 to 15 sec, CC Conc. 15.62 µmol/L, n=10, 11 | 8.3 (5.96) | 6.9 (4.66)
  0 to 15 sec, CC Conc. 31.25 µmol/L, n=10, 11 | 8.7 (6.63) | 6.0 (4.36)
  0 to 15 sec, CC Conc. 62.5 µmol/L, n=6, 10 | 8.3 (6.15) | 6.8 (3.55)
  0 to 15 sec, CC Conc. 125 µmol/L, n=5, 9 | 6.0 (1.22) | 7.1 (3.02)
  0 to 15 sec, CC Conc. 250 µmol/L, n=3, 6 | 6.3 (0.58) | 5.7 (1.21)
  0 to 15 sec, CC Conc. 500 µmol/L, n=3, 4 | 7.3 (2.52) | 7.3 (2.22)
  0 to 15 sec, CC Conc. 1000 µmol/L, n=1, 1 | 6.0 (NA) — Only one of participant analyzed at this time point. Hence SD is not calculated. | 7.0 (NA) — Only one of participant analyzed at this time point. Hence SD is not calculated.
  0 to 30 sec, CC Conc.0.49 µmol/L, n=10, 11 | 0.0 (0.00) | 0.5 (1.81)
  0 to 30 sec, CC Conc.0.97 µmol/L, n=10, 11 | 0.0 (0.00) | 0.2 (0.60)
  0 to 30 sec, CC Conc.1.95 µmol/L, n=10, 11 | 2.0 (4.64) | 1.9 (3.36)
  0 to 30 sec, CC Conc.3.9 µmol/L, n=10, 11 | 5.4 (6.59) | 4.3 (6.83)
  0 to 30 sec, CC Conc. 7.81 µmol/L, n=10, 11 | 6.7 (9.57) | 5.5 (6.42)
  0 to 30 sec, CC Conc. 15.62 µmol/L, n=10, 11 | 12.2 (9.47) | 7.5 (5.47)
  0 to 30 sec, CC Conc. 31.25 µmol/L, n=10, 11 | 11.0 (9.87) | 6.5 (5.01)
  0 to 30 sec, CC Conc. 62.5 µmol/L, n=6, 10 | 9.2 (7.19) | 7.4 (4.12)
  0 to 30 sec, CC Conc. 125 µmol/L, n=5, 9 | 6.0 (1.22) | 8.2 (4.24)
  0 to 30 sec, CC Conc. 250 µmol/L, n=3, 6 | 6.3 (0.58) | 6.7 (1.37)
  0 to 30 sec, CC Conc. 500 µmol/L, n=3, 4 | 8.7 (4.73) | 8.5 (3.51)
  0 to 30 sec, CC Conc. 1000 µmol/L, n=1, 1 | 6.0 (NA) — Only one of participant analyzed at this time point. Hence SD is not calculated. | 7.0 (NA) — Only one of participant analyzed at this time point. Hence SD is not calculated.

32. Secondary Outcome: Mean Number of Cough Counts at Each Dose of the Challenge Agent for the Citric Acid Challenge (CAC)at Visits 6 and 7 (Part C)
Description: Citric acid was administered using a dosimeter through a nebulizer pot with flow-limitation. Inhalation of increased Conc. was continued until the maximum dose was tolerated by the par. or the highest available Conc. was used. The dose-response relationship between the dose of citric acid and cough response was investigated using non-linear mixed effect modelling using Poisson and Negative Binomial distributions. When using a Poisson distribution, there was some evidence for an increase in citric acid ED50 with GSK2339345 of 41.6%, however, this was not confirmed when using a Negative Binomial distribution. The Negative Binomial distribution described the data marginally better, but the dataset was too small to make definitive conclusions. There was no treatment difference in citric acid Emax
Time Frame: After the administration of GSK2339345 or placebo (first and second 15 seconds following each dose) at Visits 6 and 7 in Part C (up to 2 weeks)
Population: CAC Population comprised of participants in the All Subjects Population for whom any CAC data were available for one or both Part C study visits. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Mean (Standard Deviation); unit: Cough count
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 9 | 9
Cough count
  0 to 15 sec, CAC Conc. 0.03 mol/L, n=9, 9 | 0.2 (0.44) | 0.2 (0.67)
  0 to 15 sec, CAC Conc. 0.06 mol/L, n=9, 9 | 0.2 (0.67) | 0.6 (1.33)
  0 to 15 sec, CAC Conc. 0.125 mol/L, n=9, 9 | 3.0 (4.66) | 1.8 (1.92)
  0 to 15 sec, CAC Conc. 0.25 mol/L, n=9, 9 | 3.7 (4.09) | 2.7 (3.43)
  0 to 15 sec, CAC Conc. 0.5 mol/L, n=9, 9 | 6.1 (5.13) | 4.3 (3.43)
  0 to 15 sec, CAC Conc. 1 mol/L, n=9, 9 | 6.0 (3.50) | 6.6 (3.40)
  0 to 15 sec, CAC Conc. 2 mol/L, n=5,7 | 5.8 (4.02) | 4.1 (3.29)
  0 to 15 sec, CAC Conc. 4 mol/L, n=5, 6 | 4.0 (3.81) | 5.3 (4.46)
  0 to 30 sec, CAC Conc. 0.03 mol/L, n=9, 9 | 0.2 (0.44) | 0.2 (0.67)
  0 to 30 sec, CAC Conc. 0.06 mol/L, n=9, 9 | 0.2 (0.67) | 0.6 (1.33)
  0 to 30 sec, CAC Conc. 0.125 mol/L, n=9, 9 | 3.2 (4.55) | 2.0 (2.06)
  0 to 30 sec, CAC Conc. 0.25 mol/L, n=9, 9 | 4.6 (6.00) | 2.7 (3.43)
  0 to 30 sec, CAC Conc. 0.5 mol/L, n=9, 9 | 7.3 (6.34) | 5.0 (4.09)
  0 to 30 sec, CAC Conc. 1 mol/L, n=9, 9 | 7.2 (4.55) | 9.3 (6.32)
  0 to 30 sec, CAC Conc. 2 mol/L, n=5, 7 | 6.8 (4.82) | 6.4 (5.32)
  0 to 30 sec, CAC Conc. 4 mol/L, n=5, 6 | 4.8 (3.83) | 6.2 (5.34)

33. Secondary Outcome: CC Agent Dose Concentration Required to Achieve C2, C5 and C6 at Visits 4 and 5 (Part B)
Description: CC was performed following the administration of GSK2339345 or placebo at Visits 4 and 5. Capsaicin was administered using a dosimeter through a nebulizer. The number of coughs in the first and second 15 sec following each dose of CC agent were recorded. Inhalation of increased conc. was continued until the maximum dose was tolerated by the participant or the highest available conc. was used. CC agent dose concentration required to achieve C2 (2 coughs were first observed [FO]), C5 (5 coughs were FO) and C6 (6 coughs were FO) are presented. All instances of missing values occurred where a participant did not achieved the required number of coughs for a parameter.
Time Frame: After the administration of GSK2339345 or placebo at Visits 4 and 5 in Part B (up to 2 weeks)
Population: CC population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the CC Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µmol/L
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 10 | 11
µmol/L
  C2, 0-15 sec, n=10, 11 | 4.181 (88.924) | 5.697 (207.575)
  C2, 0-30 sec, n=10, 11 | 4.181 (88.924) | 5.022 (194.425)
  C5, 0-15 sec, n=10, 11 | 8.967 (124.989) | 11.394 (378.087)
  C5, 0-30 sec, n=10, 11 | 8.367 (110.360) | 10.050 (535.013)
  C6, 0-15 sec, n=10, 9 | 11.834 (229.845) | 12.391 (438.063)
  C6, 0-30 sec, n=10, 10 | 10.300 (229.859) | 14.575 (908.133)

34. Secondary Outcome: CAC Agent Dose Concentration Required to Achieve C2, C5 and C6 at Visits 6 and 7 (Part C)
Description: CAC was performed following the administration of GSK2339345 or placebo at Visits 6 and 7. CA was administered using a dosimeter through a nebulizer pot with flow-limitation. Number of coughs in the first and second 15 sec following each dose of CAC agent were recorded. Inhalation of increased conc. was continued until the maximum dose was tolerated by the participants or the highest available Conc. was used. CAC agent dose concentration required to achieve C2 (2 coughs were first observed [FO]), C5 (5 coughs were FO) and C6 (6 coughs were FO) are presented. All instances of missing values occurred where a participant did not achieved the required number of coughs for a parameter.
Time Frame: After the administration of GSK2339345 or placebo at Visits 6 and 7 in Part C (up to 2 weeks)
Population: CAC population: Only those participants available at the specified time points were analyzed (represented by n=X,X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the CAC Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mol/L
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 9 | 9
mol/L
  C2, 0-15 sec, n=8, 9 | 0.209 (111.073) | 0.156 (142.342)
  C2, 0-30 sec, n=8, 9 | 0.192 (113.563) | 0.156 (142.342)
  C5, 0-15 sec, n=7, 7 | 0.305 (138.956) | 0.610 (90.153)
  C5, 0-30 sec, n=7, 8 | 0.276 (101.609) | 0.707 (127.046)
  C6, 0-15 sec, n=7, 7 | 0.371 (158.730) | 0.743 (76.173)
  C6, 0-30 sec, n= 7, 8 | 0.336 (141.375) | 0.771 (98.463)

35. Secondary Outcome: CC Agent Imputed Dose Concentration Required to Achieve C2, C5 and C6 at Visits 4 and 5 (Part B)
Description: CC was performed following the administration of GSK2339345 or placebo at Visits 4 and 5. Capsaicin was administered using a dosimeter through a nebulizer. The number of coughs in the first and second 15 sec following each dose of CC agent were recorded. Inhalation of increased Conc. was continued until the maximum dose was tolerated by the participant or the highest available Conc. was used. CC agent imputed dose concentration required to achieve C2 (at which 2 coughs were first observed [FO]), C5 (at which 5 coughs were FO) and C6 (at which 6 coughs were FO) are presented. For participants who did not complete the challenge and not reached the endpoint, values were imputed to the next dose in the challenge sequence after stopping. For participants who completed the challenge and had not reached the endpoint, values were imputed to 2000 (=twice the highest dose of capsaicin).
Time Frame: After the administration of GSK2339345 or placebo at Visits 4 and 5 in Part B (up to 2 weeks)
Population: CC Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µmol/L
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 10 | 11
µmol/L
  C2, 0-15 sec | 4.181 (88.924) | 5.697 (207.575)
  C2, 0-30 sec | 4.181 (88.924) | 5.022 (194.425)
  C5, 0-15 sec | 8.967 (124.989) | 11.394 (378.087)
  C5, 0-30 sec | 8.367 (110.360) | 10.050 (535.013)
  C6, 0-15 sec | 11.834 (229.845) | 25.850 (1279.694)
  C6, 0-30 sec | 10.300 (229.859) | 20.100 (1288.571)

36. Secondary Outcome: CAC Agent Imputed Dose Concentration Required to Achieve C2, C5 and C6 at Visits 6 and 7 (Part C)
Description: CAC was performed following the administration of GSK2339345 or placebo at Visits 6 and 7. CA was administered using a dosimeter through a nebulizer pot with flow-limitation. Number of coughs in the first and second 15 sec following each dose of CAC agent were recorded. Inhalation of increased Conc. was continued until the maximum dose was tolerated by the participants or the highest available Conc. was used. CAC agent imputed dose concentration required to achieve C2 (at which 2 coughs were first observed [FO]), C5 (at which 5 coughs were FO) and C6 (at which 6 coughs were FO) are presented. For participants who did not complete the challenge and not reached the endpoint, values were imputed to the next dose in the challenge sequence after stopping. For participants who completed the challenge and had not reached the endpoint, values were imputed to 2000 (=twice the highest dose of CA).
Time Frame: After the administration of GSK2339345 or placebo at Visits 6 and 7 in Part C (up to 2 weeks)
Population: CAC Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mol/L
Arm/Group | Placebo | GSK2339345 1000 µg
Number analyzed (Participants) | 9 | 9
mol/L
  C2, 0-15 sec | 0.314 (279.912) | 0.156 (142.342)
  C2, 0-30 sec | 0.290 (294.833) | 0.156 (142.342)
  C5, 0-15 sec | 0.630 (410.643) | 1.080 (216.073)
  C5, 0-30 sec | 0.583 (379.787) | 0.926 (185.962)
  C6, 0-15 sec | 0.735 (387.993) | 1.260 (179.623)
  C6, 0-30 sec | 0.680 (387.993) | 1.000 (152.443)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study treatment until follow-up (up to 8 weeks).
Description: SAEs and non-serious AEs were collected in participants of the All Subjects Population, comprised of all participants who received at least one dose of study medication.
Arm/Group | Placebo | GSK2339345 1000 µg
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 10/16 | 5/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | GSK2339345 1000 µg (N=14)
Tongue disclouration (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
QRS axis abnormal (Investigations) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
Hypoaesthesia oral (Nervous system disorders) | 1 | 0
Paraesthesia oral (Nervous system disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.